CLINICAL TRIAL: NCT01966510
Title: A Prospective Phase II Study to Evaluate Cord Blood Transplantation in Patients With Advanced Lymphoid Malignancies.
Brief Title: Cord Blood Transplantation in Patients With Advanced Lymphoid Malignancies
Acronym: LYMPHCORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110145
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Patients With Advanced Lymphoid Malignancies in the Absence of an HLA Identical or Mismatch Donor
Keywords: cord blood transplant; advanced lymphoid malignancies
MeSH Terms: interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cord blood transplantation (Experimental): Two cord blood units containing both together more than 3x10^7 frozen nucleated cells/Kg with no more than 2 out of 6 HLA mismatches between them and with the patients.
  Interventions: Other: Cord Blood Transplantation

INTERVENTIONS:
Other: Cord Blood Transplantation

SUMMARY:
Indication: Patients with advanced lymphoid malignancies in the absence of an HLA identical or mismatch donor.

Objectives: Overall survival at one year. Efficacy >60%, rejection rate <20%. Inclusion criteria: Age: 18-65 years old, no sibling or unrelated donor identified, low grade non-hodgkin lymphoma in third line (who already received at least one autologous transplantation); hodgkin lymphoma in early relapse (<1 year), who received at least one autologous transplantation and sensible to chemotherapy and CLL with 17p deletion or in relapse less than 2 year after a fludarabine nbased regimen or in relapse after one autologous transplantation.

Stem cell source: Two cord blood units containing both together more than 3x107 frozen nucleated cells/Kg with no more than 2 out of 6 HLA mismatches between them and with the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old
* no sibling or unrelated donor identified (9/10 or 10/10)
* with either one of these advanced lymphoid malignancies

  1. low grade non-hodgkin lymphoma in third line (who already received at least one autologous transplantation)
  2. hodgkin lymphoma in early relapse (<1 year)who received at least one autologous transplantation and sensible to chemotherapy
  3. CLL with 17p deletion or in relapse less than 2 year after a fludarabine nbased regimen or in relapse after one autologous transplantation.

Exclusion Criteria:

* No patient signed consent
* Previous allograft
* Psychiatric conditions
* HIV positive
* HVC hepatitis requiring treatment
* Previous total body irradiation (TBI)
* Any contraindication to TBI
* Any contraindication to allograft, such as cardiovascular, respiratory, renla or liver dysfunctions
* No Health care insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Engraftment | 100 days
  Neutrophils > 500/mm3 and platelets > 20 Giga/L
Chimerism | D15, D30, D60, D100, M6, M12 and M24
  using PCR
Acute Graft versus host disease (GvHD) | 100 days
Chronic graft versus host disease (GVHD) | within 2 years after inclusion
Immunologic reconstitution | D30, D60, D100, M6, M12 and M24
  phenotypic measurements of lymphocyrtes populations (T, B and NK)
Incidence of severe infectious complications | D100 and M12
  defined using criteria from EBMT (Cordonnier, www.ebmt.org)
Relapse rate | within the 2 years after inclusion
Relapse free survival | 2 years
toxicity | 2 years
  recorded according to OMS grading scale

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France